CLINICAL TRIAL: NCT03530683
Title: A Phase 1a/1b Dose-Escalation and Expansion Trial of TTI-622 in Patients With Advanced Hematologic Malignancies, Including Lymphoma, Leukemia, and Multiple Myeloma
Brief Title: A Clinical Trial to Learn About the Study Medicine Called Maplirpacept (PF-07901801), Alone and When Used in Combination With Other Medicines to Treat Participants With Advanced Hematological Malignancies, Including Lymphoma, Leukemia and Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: A business decision was made by Pfizer to terminate the study. Termination was not due to any safety concerns, requests from regulatory authorities, changes to the benefit/risk profile or any new concerns regarding the investigational product.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TTI-622-01; C4971001 (Other: Alias Study Number)
Record Dates: First submitted 2018-05-08; First posted 2018-05-21 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Lymphoma; Multiple Myeloma; Acute Myeloid Leukemia; Diffuse Large B-Cell Lymphoma
Keywords: Neoplasms; Lymphoma; Myeloma; Leukemia
MeSH Terms: conditions — Lymphoma; Multiple Myeloma; Leukemia, Myeloid, Acute; Lymphoma, Large B-Cell, Diffuse; Neoplasms; Neoplasms, Plasma Cell; Leukemia | interventions — Azacitidine; venetoclax; carfilzomib; Dexamethasone; Rituximab; isatuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- maplirpacept (PF-07901801) Monotherapy (Experimental): In the phase 1a dose- escalation part for single-agent maplirpacept (PF-07901801), participants with Relapsing or Refractory (R/R) lymphoma will be enrolled in sequential dose cohorts to receive maplirpacept (PF-07901801) QW to characterize safety, tolerability, and PK; to determine the Maximum Tolerated Dose (MTD) or P1b Starting Dose (a dose lower than or equal to the single-agent MTD), and to gain preliminary evidence of antitumor activity.
  In addition, participants with R/R Lymphoma may also be enrolled in a cohort to receive maplirpacept (PF-07901801) Q2W and a cohort to receive maplirpacept (PF-07901801) Q3W to characterize safety, tolerability, and PK; to determine the MTD; and to gain preliminary evidence of antitumor activity.
  Interventions: Drug: Maplirpacept (PF-07901801)
- Cohort A: maplirpacept (PF-07901801) + Azacitidine (Experimental): Cohort A1: participants with newly diagnosed TP53-mutated Acute Myelocytic Leukemia (AML) will be treated with maplirpacept (PF-07901801) QW + azacitidine.
  Cohort A2: participants with newly diagnosed TP53-mutated AML will be treated with maplirpacept (PF-07901801) QW + azacitidine.
  Interventions: Drug: Maplirpacept (PF-07901801); Drug: Azacitidine
- Cohort B: maplirpacept (PF-07901801) + Azacitidine and Venetoclax (Experimental): Cohort B1: elderly or unfit participants with newly diagnosed TP53-wildtype AML will be treated with maplirpacept (PF-07901801) QW + azacitidine and venetoclax
  Cohort B2: elderly or unfit participants with newly diagnosed TP53-wildtype AML will be treated with maplirpacept (PF-07901801) QW + azacitidine and venetoclax.
  Interventions: Drug: Maplirpacept (PF-07901801); Drug: Azacitidine; Drug: Venetoclax
- Cohort D1 and D2: maplirpacept (PF-07901801) + an anti-CD20 targeting agent (Experimental): Cohort D1: participants with Relapsing or Recurrent (R/R) CD20+ Diffuse Large B Cell Lymphoma (DLBCL) will be treated with maplirpacept (PF-07901801) QW, then an increased dose Q3W + an anti-CD20 targeting agent.
  Cohort D2: participants with R/R CD20+ DLBCL will be treated with maplirpacept (PF-07901801) dosed QW for 4 weeks, then an increased dose Q3W + an anti-CD20 targeting agent.
  Interventions: Drug: Maplirpacept (PF-07901801); Drug: Anti-CD20 Targeting agent
- Cohort E1 and E2: single agent maplirpacept (PF-07901801) (Experimental): Cohort E1: participants with Relapsing or Recurrent (R/R) Multiple Myeloma (MM) will be treated with single agent maplirpacept (PF-07901801) QW.
  Cohort E2: participants with R/R MM will be treated with single agent maplirpacept (PF-07901801) increased dose QW.
  Interventions: Drug: Maplirpacept (PF-07901801)
- Cohort F1, F2 and F3: maplirpacept (PF-07901801) + isatuximab, carfilzomib and dexamethasone (Experimental): Cohort F1: participants with Relapsing or Recurrent (R/R) Multiple Myeloma (MM) will be treated with increasing doses of maplirpacept (PF-07901801) + isatuximab, carfilzomib and dexamethasone.
  Cohort F2: participants with R/R MM will be treated with maplirpacept (PF-07901801) QW + isatuximab, carfilzomib and dexamethasone.
  Cohort F3: participants with R/R MM will be treated with maplirpacept (PF-07901801) increased dose QW + isatuximab, carfilzomib and dexamethasone.
  Interventions: Drug: Maplirpacept (PF-07901801); Drug: Carfilzomib; Drug: Dexamethasone; Drug: Isatuximab
- Cohort C1, C2 and C3: maplirpacept (PF-07901801) + Carfilzomib and Dexamethasone (Experimental): Cohort C1: participants with Relapsing or Refractory (R/R) Multiple Myeloma (MM) will be treated with maplirpacept (PF-07901801) QW
  + carfilzomib and dexamethasone.
  Cohort C2: participants with R/R MM will be treated with maplirpacept (PF-07901801) QW + carfilzomib and dexamethasone.
  Cohort C3: participants with R/R MM will be treated with maplirpacept (PF-07901801) Q2W + carfilzomib and dexamethasone.
  Interventions: Drug: Maplirpacept (PF-07901801); Drug: Carfilzomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Maplirpacept (PF-07901801) — maplirpacept (PF-07901801) will be administered by intravenous infusion at ranging doses, as determined from sequential dosing cohorts.
  Other Names: SIRPα-IgG4 Fc; TTI-622
Drug: Azacitidine — intravenous (IV) or subcutaneous (SC) daily for 7 days, repeated every 4 weeks
  Other Names: VIDAZA
  Arms: Cohort A: maplirpacept (PF-07901801) + Azacitidine; Cohort B: maplirpacept (PF-07901801) + Azacitidine and Venetoclax
Drug: Venetoclax — orally daily for each day of each cycle (first 7 doses taken in clinic). The ramp-up and target dose of venetoclax will be adjusted per the package insert in subjects who are taking concomitant moderate or strong CYP3A4 inhibitors or posaconazole
  Other Names: VENCLEXTA
  Arms: Cohort B: maplirpacept (PF-07901801) + Azacitidine and Venetoclax
Drug: Carfilzomib — Days 1, 8, and 15 of 28-day cycles; starting dose IV given on Cycle (C) 1 Day (D) 1, and if tolerated, then increased dose via IV given starting on C1D8 and subsequent doses thereafter.
  Other Names: KYPROLIS
  Arms: Cohort C1, C2 and C3: maplirpacept (PF-07901801) + Carfilzomib and Dexamethasone; Cohort F1, F2 and F3: maplirpacept (PF-07901801) + isatuximab, carfilzomib and dexamethasone
Drug: Dexamethasone — starting dose via IV on Days 1, 8, 15, and increased dose via IV on 28-day cycles
  Arms: Cohort C1, C2 and C3: maplirpacept (PF-07901801) + Carfilzomib and Dexamethasone; Cohort F1, F2 and F3: maplirpacept (PF-07901801) + isatuximab, carfilzomib and dexamethasone
Drug: Anti-CD20 Targeting agent — Days 1,8,15, and 22 of the first 28-day cycle and then on Day 1 of subsequent 21-day cycles. The anti-CD20 targeting agent will be administered for a total of eight doses, and then Cohort F1, F2 and F3: TTI-622 + isatuximab, carfilzomib and dexamethasone Cohort C1, C2 and C3: TTI-622 + Carfilzomib and Dexamethasone will be continued as single-agent therapy.
  Other Names: Ruxience or Rituxan
  Arms: Cohort D1 and D2: maplirpacept (PF-07901801) + an anti-CD20 targeting agent
Drug: Isatuximab — F1: IV dose C0D1, C0D8, C0D15 and C0D22 (lead in phase);weekly during Cycle 1; Cycle 2 and beyond will be administered on Days 1 and 15 (Q2W).
  F2 and F3: IV dose C0D1 and C0D8 (lead in phase); C1D1, C1D8, C1D15 and C1D22; Cycle 2 and beyond will be administered on days 1 and 15 (Q2W). Carfilzomib: IV dose on days 1 and 2 of cycle 1; then increased IV dose on days 8, 9, 15, and 16 of cycle 1; cycle 2 and beyond: increased IV dose on days 1, 2, 8, 9, 15, and 16. Dexamethasone IV or PO on days 1, 2, 8, 9, 15, 16, 22, and 23 starting cycle 1.
  Other Names: Sarclisa
  Arms: Cohort F1, F2 and F3: maplirpacept (PF-07901801) + isatuximab, carfilzomib and dexamethasone

SUMMARY:
The purpose of this clinical trial is to learn how the experimental medicine maplirpacept (PF-07901801) affects people with various types of blood cancers:

* relapsed or refractory (R/R) lymphoma
* multiple myeloma
* newly diagnosed acute myeloid leukemia (AML).

This trial will be conducted in the outpatient setting in 2 parts, phase 1a and phase 1b. You may only participate in one part of the study.

During phase 1a of this study, we will explore how much maplirpacept (PF-07901801), when used by itself, can be safely used.

If you have lymphoma, the study medicine maplirpacept (PF-07901801) will be given by infusion through a vein once a week or once every 2 weeks or every 3 weeks as determined by your doctor. Following your first dose, you will be expected to come back twice more the first week. From week 2, you will have weekly visits for blood tests, questions about your medications, any side effects, or illnesses you may have experienced and your cancer response. After you have completed 21 days (for every week dosing) or 42 days (for every 2- or 3-weeks dosing), your doctor will discuss whether you should stop study treatment or continue.

If you continue, you will be expected to come back weekly for blood tests, vital signs, a brief physical exam, asked about any side effects or illnesses you may have experienced and medications you may be taking. The dosing schedule you are assigned to will continue until your disease has worsened, significant side effects occur or other reasons that lead you and your doctor to decide treatment may be stopped.

To be eligible for the first part of the study you must be 18 years or older, your disease has worsened after receiving other medicines approved for blood cancer, no other treatment options exist for you, a sample of your tissue for exploratory research which can be taken from tissue already obtained or if necessary, a new sample of your tissue will be taken so your disease may be seen and measured on routine tests/scans. If you have had radiation therapy or received any anticancer medication within 14 days before the planned start of study treatment your doctor will let you know if you are eligible to participate in the study. If you have had major surgery within 30 days before the planned start of study treatment you may not be eligible to participate.

The phase 1a part of the study may last up to 51/2 years. How long you participate in this study depends on side effects you may have to the study drug. It also depends on how your cancer responds to the study drug. Therefore, you may remain in the study as long as you and your study doctor think you may benefit. However, you are free to stop taking part in this study at any time and for any reason.

During phase 1b part of this study, we will explore how much maplirpacept (PF-07901801), when used with other anticancer medicine(s), can be safe and reduce cancer growth. In the phase 1b part of this study, you will receive maplirpacept (PF-07901801) and other anticancer medicine(s). Which medicine combination you will receive depends on the types of cancer under treatment. Your treatment experiences will be examined to determine if maplirpacept (PF-07901801) when given with other anticancer medicine(s), is safe and can reduce cancer growth.

To be eligible for the second part of the study you may have newly diagnosed Acute Myelocytic Leukemia with or without a genetic mutation or you have Multiple Myeloma or Diffuse Large B Cell Lymphoma, and your disease has worsened.

The Phase 1b part of this study may last as long as you and your study doctor think you may benefit which could be up to approximately 31/2 years. How long you participate in this study depends on side effects you may have to the study drug. It also depends on how your cancer responds to the study drug. Therefore, you may remain in the study as long as you and your study doctor think you may benefit. However, you are free to stop taking part in this study at any time and for any reason.

DETAILED DESCRIPTION:
This is a trial of maplirpacept (PF-07901801) in subjects with relapsed or refractory lymphoma or multiple myeloma (MM) and subjects with newly diagnosed acute myeloid leukemia (AML).

This trial will be conducted in 2 phases: Phase 1a (Dose-Escalation Phase for Single-Agent maplirpacept (PF-07901801) and Phase 1b maplirpacept (PF-07901801) Combinations and Single-Agent.

In the Dose-Escalation Phase for Single-Agent maplirpacept (PF-07901801), subjects with relapsed or refractory lymphoma will be enrolled in sequential dose cohorts.

In the Combination and Single-Agent Treatment part, subjects will be included in 1 of 14 cohorts: (Cohort A1 and A2) subjects with newly diagnosed TP53-mutated AML will be treated with maplirpacept (PF-07901801) + azacitidine; (Cohort B1 and B2) elderly subjects or subjects unfit for intensive induction chemotherapies with newly diagnosed TP53-wildtype AML will be treated with maplirpacept (PF-07901801) + azacitidine and venetoclax; (Cohort C1, C2, and C3) subjects with relapsed or refractory MM will be treated with maplirpacept (PF-07901801) + carfilzomib and dexamethasone;(Cohort D1 and D2) subjects in relapsed or refractory CD20+ diffuse large B-cell lymphoma will be treated with maplirpacept (PF-07901801) + an anti-CD20 targeting agent; (Cohort E1 and E2) subjects with relapsed refractory MM will be treated with single-agent maplirpacept (PF-07901801); and (Cohorts F1, F2 and F3) with relapsing or refractory MM will be treated with increasing doses of maplirpacept (PF-07901801) + isatuximab, carfilzomib and dexamethasone.

ELIGIBILITY:
Key Inclusion Criteria (Phase 1a and Phase 1b, all Cohorts):

1. Available fresh or archived tumor tissue.
2. Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2.
3. Adequate coagulation function.
4. Adequate hepatic function.
5. Adequate hematologic status.
6. Adequate renal function.
7. Recovery from non-hematopoietic toxicities of previous anticancer drugs or radiotherapy or previous surgeries to ≤Grade 1 (or to baseline grade if condition was pre-existing).

Key Inclusion Criteria (Phase 1a): Histologically confirmed relapsed/refractory, transfusion- independent lymphoma (Hodgkin or non-Hodgkin) per the 2014 Lugano classification.

Key Inclusion Criteria (Phase 1b Cohort A1 and A2): Histologically confirmed, newly diagnosed TP53-mutated Acute Myeloid Leukemia (AML).

Key Inclusion Criteria (Phase 1b Cohort B1 and B2): Histologically confirmed, newly diagnosed TP53-wildtype AML, elderly or unfit for more aggressive treatment.

Key Inclusion Criteria (Phase 1b Cohorts C1, C2, C3 and E1, E2, F1, F2, F3): Histologically documented relapsed/refractory Multiple Myeloma (MM).

Key Inclusion Criteria (Phase 1b Cohort D1 and D2): Pathologically confirmed relapsed/refractory diffuse large B-cell lymphoma (DLBCL)

Key Exclusion Criteria (Phase 1a and Phase 1b, all Cohorts):

1. Known, current central nervous system disease involvement.
2. Use of any investigational agent or any anticancer drug within 14 days before planned start of study treatment (within 4 weeks for antibody-based therapies and within 8 weeks for cell-based therapies).
3. Subjects who have undergone radiation therapy within 14 days of study treatment administration.
4. Hematopoietic stem cell transplant within 90 days before the planned start of study treatment or subjects with active graft-vs-host disease, with the exception of Grade 1 skin involvement.
5. Major surgery within 30 days before planned start of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2024-07-18 (Actual)

PRIMARY OUTCOMES:
Phase 1a: Number of adverse events (AE) by severity | Through study completion, up to 18 months
  To characterize the safety profile (incidence of AEs)
Phase 1a: Number of AEs by Frequency | Through study completion, up to 18 months
  To characterize the safety profile (incidence of AEs) and
Phase 1a: Number of participants with Dose-Limiting Toxicities (DLT) | Up to 21-42 days
  To characterize the dose limiting toxicities (DLTs) of TTI-622.
Phase 1b: Number of adverse events (AE) by severity | Through study completion, up to 30 months
  To characterize the safety profile (incidence of AEs) of TTI-622 given in combinations or as a single agent.
Phase 1b: Number of adverse events (AE) by frequency | Through study completion, up to 30 months
  To characterize the safety profile (incidence of AEs) of TTI-622 given in combination or as a single agent.
Phase 1b: Number of participants with disease response | Through study completion, up to 30 months
  To evaluate response rate of each combination treatment in the (7) combination cohorts (A1,A2, B1, B2, C1, C2, C3, D1, D2, F1, F2, F3) and for single agent treatment (Cohort E1 and E2). For AML, response = CR. For MM, response = CR+sCR+VGBR+PR. For DLBCL, OR=CR+PR
Phase 1a: Maximum Tolerated Dose (MTD) | Baseline (the start of each sequentially increased treatment dose), up to the 3rd evaluable patient completes DLT observation period of 21 or 42 days.
  To characterize the highest dose level for which no more than 1 participant in a dose cohort experienced DLTs.
Phase 1b: Recommended dose of TTI-622 in combination with selected anticancer treatments | Through study completion, up to 30 months
  To characterize the recommended dose of TTI-622 in combination with selected anticancer treatments in 5 patient populations:
  * TTI-622 plus azacitidine in newly diagnosed TP53-mutated AML
  * TTI-622 plus azacitidine and venetoclax in elderly (>/= 75 years old) or unfit, newly diagnosed TP53-wildtype AML
  * TTI-622 plus Carfilzomib and dexamethasone in Carfilzomib-refractory, Relapsed/Refractory (R/R) multiple myeloma (MM) after 3 or more prior lines of therapy
  * TTI-622 plus an anti-CD20 targeting agent (such as ruxience or rituxan) in R/R CD20+ DLBCL after 1 or more prior lines of therapy
  * TTI-622 plus isatuximab, carfilzomib and dexamethasone in R/R MM after 1-3 prior lines of therapy
Phase 1b: Recommended dose of TTI-622 as a single agent | Through study completion, up to 30 months
  To characterize the recommended dose of TTI-622 as a single agent in patients with R/R MM after 3 or more prior lines of therapy.
Number of participants with response assessments that show preliminary efficacy | Through study completion, up to 30 months
  To evaluate preliminary efficacy of each combination treatment in the selected patient populations and for single-agent treatment in R/R MM

SECONDARY OUTCOMES:
Phase 1a: TTI-622 PK parameter AUC0-t | Through study completion, up to 18 months
  To characterize AUC0-t of TTI-622.
Phase 1a: TTI-622 PK parameter Cmax | Through study completion, up to 18 months
  To characterize Cmax of TTI-622.
Phase 1a: Incidence of anti-drug antibodies (ADA) | Through study completion, up to 18 months
  To characterize the immunogenicity of TTI-622.
Phase 1a: Number of participants with overall response rate (ORR) for participants treated with TTI-622. | Through study completion, up to 18 months
  To determine the disease response.
Phase 1a: Number of participants with disease control rate (DCR) | Through study completion, up to 18 months
  To determine the disease control rate (DCR) for participants treated with TTI-622.
Phase 1a: Time to response (TTR) | Through study completion, up to 18 months
  To determine the time to response (TTR) for participants treated with TTI-622.
Phase 1a: Duration of Response (DR) | Through study completion, up to 18 months
  To determine the duration of response (DR) for participants treated with TTI-622.
Phase 1a: Progression free survival (PFS) | Through study completion, up to 18 months
  To determine the progression free survival (PFS) time for participants treated with TTI-622.
Phase 1b: TTI-622 PK parameter Cmax when combined with selected anticancer treatments or as a single agent | Through study completion, up to 30 months
  To characterize Cmax of TTI-622 when combined with selected anticancer treatments or as a single agent.
Phase 1b: incidence of anti-drug antibodies (ADA) Immunogenicity of TTI-622 when combined with selected anticancer treatments or as a single agent | Through study completion, up to 30 months
  To characterize the immunogenicity of TTI-622 when combined with selected anticancer treatments or as a single agent
Phase 1b: Number of participants with disease control rate (DCR) | Through study completion, up to 30 months
  To determine the disease control rate (DCR) for participants treated with TTI-622 when combined with selected anticancer treatments or as a single agent.
Phase 1b: Time to response (TTR) | Through study completion, up to 30 months
  To determine the time to response (TTR) for participants treated with TTI-622 when combined with selected anticancer treatments or as a single agent.
Phase 1b: Event-free survival (EFS) | Through study completion, up to 30 months
  To determine event-free survival (EFS; for Cohorts A and B) time for participants treated with TTI-622 when combined with selected anticancer treatments or as a single agent.
Phase 1b: Duration of response (DR) | Through study completion, up to 30 months
  To determine the duration of response (DOR) for participants treated with TTI-622 when combined with selected anticancer treatments or as a single agent.
Phase 1b: Progression-free survival (PFS) | Through study completion, up to 30 months
  To determine the progression-free survival (PFS) time for participants treated with TTI-622 when combined with selected anticancer treatments or as a single agent.
Phase 1b: Number of Participants With Minimal Residual Disease Burden (MRD) Positive, Negative and Not Evaluable (NE) Status | Through study completion, up to 30 months
  To determine minimal residual disease (MRD; for Cohorts A, B, C , E and F) for participants treated with TTI-622 when combined with selected anticancer treatments or as a single agent.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (62):
- United States (62):
  - Keck Hospital of USC, Los Angeles, California
  - LAC+USC Medical Center, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Keck Hospital of USC Pasadena, Pasadena, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - HealthONE Presbyterian/St. Luke's Medical Center, Denver, Colorado
  - Christiana Care Health Services, Newark, Delaware
  - Christiana Care Hematology Oncology - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants, PA, Helen F. Graham Cancer Center, Newark, Delaware
  - Christiana Care Health Services - Christiana Hospital, Newark, Delaware
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Tampa General Hospital Cancer Institute, Tampa, Florida
  - Tampa General Hospital, Tampa, Florida
  - Blood and Marrow Transplant Group of Georgia, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Indiana Blood & Marrow Transplantation, Indianapolis, Indiana
  - Indiana Blood and Marrow Transplantation-Administrative Offices, Indianapolis, Indiana
  - Indiana Blood and Marrow Transplantation-Clinic, Indianapolis, Indiana
  - Norton Cancer Institute, St Matthews Campus, Louisville, Kentucky
  - Norton Cancer Institute, St. Matthews Campus, Attn. Becky Champion, PharmD, Louisville, Kentucky
  - Norton Diagnostic Center-Dupont (PET Scans), Louisville, Kentucky
  - Norton Women & Children's Hospital, Louisville, Kentucky
  - University of Michigan Hospitals, Ann Arbor, Michigan
  - University of Michigan, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Karmanos Cancer Institute Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Memorial Sloan Kettering Cancer Center at Basking Ridge, Basking Ridge, New Jersey
  - Summit Medical Group Cancer Center, Florham Park, New Jersey
  - Memorial Sloan Kettering Cancer Center at Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center at Montvale, Montvale, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center at Commack, Commack, New York
  - Memorial Sloan Kettering Cancer Center at Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center - Investigational Drug Service Pharmacy, Long Island City, New York
  - Memorial Sloan Kettering Cancer Center - David H. Koch Center, New York, New York
  - Memorial Sloan Kettering Cancer Center (Outpatient Center), New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Memorial Sloan Kettering Cancer Center at Nassau, Uniondale, New York
  - Novant Health Cancer Institute - Research Office, Charlotte, North Carolina
  - Novant Health Cancer Institute Hematology - Charlotte, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Novant Health Cancer Institute - Research Office, Winston-Salem, North Carolina
  - Novant Health Cancer Institute Hematology - Forsyth, Winston-Salem, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Gabrail Cancer Center Research, Canton, Ohio
  - Sidney Kimmel Cancer Center, Clinical Trials Organization, Philadelphia, Pennsylvania
  - Sidney Kimmel Cancer Center, Research Support Services, Philadelphia, Pennsylvania
  - Thomas Jefferson University - Clinical Research Institute, Philadelphia, Pennsylvania
  - Thomas Jefferson University Investigational Drug Services, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Investigational Drug Service, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Medical Oncology, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - Prisma Health, Institute for Translational Oncology Research, Clinical Research Unit, Greenville, South Carolina
  - Prisma Health-Upstate Cancer Institute, Greenville, South Carolina
  - University of TN Medical Center, Knoxville, Tennessee
  - Oncology Consultants P.A., Houston, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Swedish Cancer Institute, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=TTI-622-01